CLINICAL TRIAL: NCT06675357
Title: Novel FAP-targeted Approach to Imaging Patients With or High-risk for Metastatic Prostate Cancer
Brief Title: Using FAPI PET/MRI to Evaluate Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-0747; A539300 (Other: UW Madison); Protocol Version 8/4/25 (Other: UW Madison); UW24045 (Other: UWCCC OnCore ID); Prostate SPORE (Other: UW Madison)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Metastatic Disease; Prostate Cancers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Fibroblast activation protein inhibitor (FAPI) (Experimental): FAPI radiotracer will be used during PET
  Interventions: Radiation: FAPI; Procedure: Positron Emission Tomography (PET); Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: FAPI — 5 +/- 2 mCi of Ga-FAPI-46
Procedure: Positron Emission Tomography (PET) — Undergo PET scan
Procedure: Magnetic Resonance Imaging — Undergo MRI scan

SUMMARY:
The goal of this clinical trial is to gain more information about how FAPI (fibroblast activation protein inhibitor) binds to certain type of cells in the tumor tissue. The main question it aims to answer is how this information can be used to better diagnose and track prostate cancer.

Participants will undergo two PET/MRI scans during two research visits, each of which may last up to 2.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able and willing to provide informed consent
* Known diagnosis of prostate cancer
* Scheduled for or recently performed (within 4 weeks) standard-of-care PSMA PET
* Optional: Scheduled for SOC biopsy of an established or suspected non-osseous, non-nodal metastases.
* Willing and able to undergo PET/MRI as part of this research

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Contraindication(s) to or inability to undergo PET/MRI
* Participants for whom PET/MRI will delay timely delivery of treatment
* Participants requiring intravenous (IV) conscious sedation for imaging care; those requiring mild, oral anxiolytics for the clinical MRI will be allowed to participate as long as the following criteria are met:
* Have their own prescription for the medication
* The informed consent process is conducted prior to the self-administration of this medication
* Come to the research visit with a driver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Performance of FAPI for lesion detection | Duration of scan, up to 80 minutes
  Sensitivity and specificity for lesion detection on FAPI will be compared with that of PSMA PET, using a composite reference standard (all available histology, follow up clinical/standard of care imaging, serum PSA).
Lesion FAPI uptake on PET | Duration of scan, up to 80 minutes
  FAPI uptake as measured by SUV will be correlated against tissue FAP positivity on immunohistochemistry and FAP expression on qPCR, using linear regression.
Total FAPI-positive tumor volume change | Duration of scan, up to 80 minutes
  The total FAPI-positive tumor volume between pre- and post-treatment exams will be measured and compared to PSMA-response, other standard-of-care imaging response, and overall survival when available, using odds ratios for treatment response and Kaplan-Meier curve for survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Pirasteh, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data with GE Healthcare: images, diagnosis, image quality scores, quantitative PET/MR measurements, BMI, weight, height, age and gender. The Department of Radiology Medical Imaging Research Support (MIRS) Radius team will serve as an honest broker for the sharing of de-identified data.